CLINICAL TRIAL: NCT00821548
Title: Electrostimulation of Shoulder Girdle and Quadriceps Muscles in Facioscapulohumeral Muscular Dystrophy Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Centre Hospitalier Universitaire de Nice - Estelle MARTINEZ
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 07-CIR-01
Record Dates: First submitted 2009-01-12; First posted 2009-01-13 (Estimated); Last update posted 2009-01-13 (Estimated); Status verified 2009-01

CONDITIONS: Facioscapulohumeral Muscular Dystrophy
Keywords: facioscapulohumeral muscular dystrophy; electrostimulation; training
MeSH Terms: conditions — Muscular Dystrophy, Facioscapulohumeral | interventions — Transcutaneous Electric Nerve Stimulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): Electrostimulation of the muscles of the scapular belt and the femoris quadristocks
  Interventions: Procedure: electrostimulation

INTERVENTIONS:
Procedure: electrostimulation — Electrostimulation of shoulder girdle and quadriceps muscles in facioscapulohumeral muscular dystrophy patients

SUMMARY:
The investigators evaluated clinical tolerance, biological tolerance, feasibility and efficacy of daily electrostimulation training of shoulder girdle and quadriceps muscles in 10 patients with facioscapulohumeral muscular dystrophy, the third most common inherited myopathy.

DETAILED DESCRIPTION:
Autosomal dominant FSHD is characterized by selective pattern of muscle involvement. Weakness and atrophy typically involve facial and shoulder girdle muscles, and progressively anterior forearm and foreleg muscles and pelvic girdle muscles.

The physiopatholgical mechanism of this disease, due to a deletion of repeated units named D4Z4 located on 4q35, is still controversial. Up to date, no curative therapy is available for these patients. We proposed in the present study to test feasibility, clinical and biological tolerance and efficacy of shoulder muscle training by electrostimulation in a group of FSHD patients. 10 patients displaying classical FSHD phenotype participate to this study consisting in daily session of shoulder girdle and quadriceps muscles electrostimulation of 23 minutes for a period of 5 months.

We evaluated: clinical tolerance by daily pain and fatigue analogic scales, biological tolerance by measuring CK; feasibility: by measuring the monthly score of participation to sessions; the efficacy by manual muscle testing, quantitative muscle assessment, fatigue severity scale.

ELIGIBILITY:
Inclusion Criteria:

* 18 to 75 years old patient
* FSHD diagnosis confirmed by molecular biology
* FSHD clinical phenotype including shoulder girdle and quadriceps involvement
* Patient with Vignos scale ≤ 5 (patient able to walk)
* Patient with health insurance
* Patient that could be followed for at least 6 months

Exclusion Criteria:

* Patient with monolateral or bilateral scapular omopexia
* Patient that has already had electrostimulation training
* Patients with CK values > 5 time normal values
* Patient that has not signed informed consent
* Patient with cancer, collagenopathies or others joint diseases
* Pregnancy and breast-feeding
* Patient on guardianship or trusteeship.
* Patient actively participating to other biomedical researches or whose exclusion period is not ended
* Patient with a formal contraindication to the protocol detected by inclusion examinations

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2008-01; Primary Completion 2008-07 (Actual); Study Completion 2008-07 (Actual)

PRIMARY OUTCOMES:
Clinical tolerance evaluated by fatigue and pain analogic scale. Biological tolerance:evaluated by measuring CK values.The feasibility:evaluated by considering monthly average length of sessions, monthly score of participation to sessions | daily, 1, 3 and 5 months

SECONDARY OUTCOMES:
Efficacy of electrostimulation training in FSHD patients will be evaluated comparing manual muscle testing, Barré test, quantitative muscle assessment, fatigue severity scale, 6 minutes walking test before the therapy | after 3 months of therapy and at the end of the study, after 5 months.

CONTACTS AND LOCATIONS:
Locations (1):
- CHU de Nice, Nice, France

REFERENCES:
- [Derived] Colson SS, Benchortane M, Tanant V, Faghan JP, Fournier-Mehouas M, Benaim C, Desnuelle C, Sacconi S. Neuromuscular electrical stimulation training: a safe and effective treatment for facioscapulohumeral muscular dystrophy patients. Arch Phys Med Rehabil. 2010 May;91(5):697-702. doi: 10.1016/j.apmr.2010.01.019. PMID 20434605